CLINICAL TRIAL: NCT01598272
Title: A Phase IV, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Single-Center Study on the Effects of a Proprietary Blend of Herbal Extract Supplement on Cellular Detoxification, Inflammation, and Cumulative Cognitive Index as Well as Gene Expression in Middle-Aged Adult Women.
Brief Title: Effects of a Proprietary Blend of Herbal Extract Supplement on Cellular Detoxification, Inflammation, and Cumulative Cognitive Index as Well as Gene Expression in Middle-Aged Adult Women
Acronym: Pharmanex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: Aspen Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11-PHX-03-NU-01
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Anti Aging
Keywords: Ginseng; Cordyceps; Pomegranate; Red Orange; Grape Seed; Broccoli Seed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitality product AM + Vitality product PM (Experimental): Dietary Supplement:
  Proprietary blend of ginseng, cordyceps, and pomegranate + proprietary blend of broccoli seed, red orange, and grape seed taken twice a day for 8 weeks.
  Interventions: Dietary Supplement: Vitality product AM + Vitality product PM
- Placebo (Placebo Comparator): Dietary Supplement: Placebo Placebo taken twice a day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitality product AM + Vitality product PM — Vitality AM: Tak 6 capsules daily for 56 days Vitality PM: Take 2 capsules daily for 56 days
  Arms: Vitality product AM + Vitality product PM
Dietary Supplement: Placebo — Placebo AM: Take 6 capsules daily for 56 days Placebo PM: Take 2 capsules daily for 56 days
  Arms: Placebo

SUMMARY:
Determine the effects of 8 week Investigational Supplement on cellular detoxification and gene expression profiles

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 35-73 years
2. Signed informed consent
3. BMI between 23 and 35 kg/m2
4. A resting normotensive blood pressure is defined as a systolic blood pressure between 90-145 mmHg and a diastolic blood pressure of 50 90 mmHg
5. BioPhotonic scanner score below 30,000
6. Use of effective method of contraception by females of childbearing [potential and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study]. Acceptable methods of contraception include oral, injectable, or implantable contraceptives; intrauterine devices, diaphragm plus spermicide; or any double barrier method. Women who have had a hysterectomy or tubal ligation at least 6 months prior to Visit 1 or who have been post-menopausal for at least 1 year prior to Visit 1 are not considered to be of childbearing potential.
7. Ability to speak and understand English.
8. Willing to consume one high-fat high carbohydrate meal at the last visit consisting of 1 McDonald's egg Mcmuffin with cheese (no meat), 1 Sausage McMuffin with cheese (no egg), 2 hashbrowns, 1 12 oz Coke Cola or Sprite.
9. Willing to not exercise the morning of your last visit

Exclusion Criteria:

1. Self-reported chronic condition that may affect subject safety (e.g., diabetes, cardiovascular disease) or significantly impact product effectiveness (e.g., chronic fatigue)
2. Pregnancy/suspected pregnancy, breastfeeding or planning to become pregnant during the course of the study.
3. Antihypertensive medication use.
4. Allergies to any ingredients contained in the Investigational Product.
5. Consumption of more than 600 mg of caffeine from all sources per day (equivalent to 24 oz. caffeinated coffee, 96 oz. of soda, 60 oz. of tea, 60 oz. energy drinks , or a combination thereof).
6. Consumption of herbal supplement known to affect energy levels (e.g., ginseng, cordyceps, licorice, Lycium, pomegranate, etc.).
7. Consumption of any of the supplements included in the formulas (Cordyceps sinensis, Panax Ginseng extract, pomegranate extract, red orange complex, grape seed extract or broccoli seed extract).
8. Known iron deficiency anemia.
9. Treatment for insomnia or depression within 30-days prior to the screening visit.
10. Recently started taking medication known to effect energy (e.g., thyroid medication). If taking medication (e.g., thyroid medication), must be stable for at least four months.
11. Tobacco (e.g. cigarettes, chewing tobacco, pipe, nicotine patches) use within 30-days prior to the screening visit.
12. Planned surgical procedure during the course of the study.
13. Currently participating in another study or have done so within 30 days prior to the screening visit or is likely to enroll in another clinical or nutritional study.
14. Any laboratory value that the investigator deems clinically significant.
15. Currently participating in a weight loss program or planning to go on a weight loss diet during the course of the study.
16. Allergies to egg or dairy products, Vegetarian or unwilling to consuming sausage.

Ages: 35 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Determine effects of investigational supplement on gene expression profiles. | Day 0, Day 28, Day 56
  Gene Expression Panel (microarray PBMCs), Inflammatory Panel, Oxidative stress Markers-including glutathione panel and F2 isoprostane, Anti-oxidant panel, and Lipid Panel

SECONDARY OUTCOMES:
Establish a safety profile of investigational supplement | Day 0, Day 28, Day 56
  Measure number of participants with adverse events. Fasted Safety Labs (chemistry, hematology, Coagulation)compared to baseline.
Determine effects of investigational supplement on markers of inflammation | Day 0, Day 28, Day 56
Determine effects of investigational supplement on composite cognitive index | Day 0, Day 28, Day 56
Determine changes in scoring on HADS assessment (Hospital Anxiety & Depression Scale) | Day 0, Day 28, Day 56
  Questionnaire: Hospital Anxiety and Depression Scale (HADS)
Determine changes in Quality of Life | Day 0, Day 28, Day 56
  SF-36 (Quality of Life Assessment)
Determine changes in sleep patterns and quality | Day 0, Day 28, Day 56
  Sleep measurement scale.
Determine changes to overall health | Day 0, Day 28, Day 56
  Abbreviated Physical Exam
Determine changes to biological age scanning (Digital Pulse Wave Analyzer (DPA) | Day 0, Day 28, Day 56
  Digital Pulse Wave Analyzer
Determine changes in Biophotonic Scanner Scores | Day 0, Day 28, Day 56
  Measure antioxidants in the palm of the skin.
Determine changes in skin advanced glycation endproducts (AGE) levels | Day 0, Day 28, Day 56
  AGE Reader

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris, DO, Principal Investigator — Aspen Clinical Research
Locations (1):
- Aspen Clinical Research, Orem, Utah, United States